CLINICAL TRIAL: NCT00750555
Title: Phase II Study of Maintenance of Tarceva (Erlotinib) in Patients With Locally Advanced Head and Neck Cancer
Brief Title: Maintenance of Tarceva (Erlotinib) in Patients With Locally Advanced Head and Neck Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI Law left Geisinger-study terminated prematurely - 4 patients enrolled
Sponsor: Geisinger Clinic (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0153; OSI4178S
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Head and Neck Cancer
Keywords: squamous cell cancer of head and neck; SCCHN
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — 150 mg per day orally until disease progression occurs, up to a maximum of 12 months
  Other Names: Tarceva

SUMMARY:
Phase II Study of Maintenance Tarceva (Erlotinib) in patients with locally advanced Head and Neck Cancer after treatment with curative intent

ELIGIBILITY:
Inclusion Criteria:

* Stage III, IV SCCHN
* Completed curative treatment

Exclusion Criteria:

* Prior chemotherapy or radiotherapy
* Recurrent disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Law, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Health System, Danville, Pennsylvania, United States

REFERENCES:
- See also: Click here for more information about Geisinger Health System — http://www.geisinger.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After the enrollment of 4 participants in this study, the PI left Geisinger. Geisinger does not have any details regarding which Arm/Group participants were assigned to.
Groups:
- One Year Disease Free: Erlotinib: 150 mg per day orally until disease progression occurs, up to a maximum of 12 months
Period: Overall Study
Arm/Group | One Year Disease Free
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Per our current document retention policy, and the fact that the investigator, study staff, and record owner are no longer employed at our site, we do not have any collected data for baseline analysis population.
Arm/Group | One Year Disease Free
Number analyzed (Participants) | 0
Age, Categorical
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: One Year Disease Free
Description: Per our current document retention policy, and the fact that the investigator, study staff, and record owner are no longer employed at our site, we do not have any collected data for pre-specified Primary and Secondary Outcome Measures to report in Outcome Measure data table.
Time Frame: 1 year
Population: Per our current document retention policy, and the fact that the investigator, study staff, and record owner are no longer employed at our site, we do not have any collected data for pre-specified Primary and Secondary Outcome Measures to report in Outcome Measure data tables.
Arm/Group | One Year Disease Free
Number analyzed (Participants) | 0

2. Secondary Outcome: Overall Survival
Description: Per our current document retention policy, and the fact that the investigator, study staff, and record owner are no longer employed at our site, we do not have any collected data for pre-specified Primary and Secondary Outcome Measures to report in Outcome Measure data tables.
Time Frame: 2 years
Population: as for outcome 1
Groups:
- Overall Survival: Erlotinib: 150 mg per day orally until disease progression occurs, up to a maximum of 12 months
Arm/Group | Overall Survival
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Per our current document retention policy, and the fact that the investigator, study staff, and record owner are no longer employed at our site, we do not have any collected data to report in Adverse Events.
Arm/Group | One Year Disease Free
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No